CLINICAL TRIAL: NCT00994045
Title: Coagulopathy During Surgery for the Repair of Extent 4 Thoraco-Abdominal Aortic Aneurysms - Feasibility Study of the Use of Fibrinogen Concentrate by Infusion in Place of Fresh Frozen Plasma.
Brief Title: Fibrinogen as an Alternative to FFP in Aortic Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); CSL Behring (Industry)
Responsible Party: Principal Investigator, Alastair Nimmo, Dr, University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIB692; EudraCT 2009-016709-41
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Coagulopathy in Patients Having Thoraco-Abdominal Aneurysm Repair
Keywords: Thoraco-Abdominal Aneurysm (TAAA); Coagulopathy; Fresh Frozen Plasma; Fibrinogen Concentrate
MeSH Terms: conditions — Hemostatic Disorders | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh Frozen Plasma (Active Comparator)
  Interventions: Biological: Fresh Frozen Plasma
- Fibrinogen concentrate (Experimental)
  Interventions: Biological: Fibrinogen concentrate

INTERVENTIONS:
Biological: Fibrinogen concentrate — Fibrinogen concentrate will be administered initially at 2 grammes per hour by continuous infusion. This rate will be adjusted in response to the clinical picture and results of point of care coagulation tests. The infusion will be used intra-operatively.
  Other Names: Haemocomplettan P; ATC code: B02B B01
  Arms: Fibrinogen concentrate
Biological: Fresh Frozen Plasma
  Arms: Fresh Frozen Plasma

SUMMARY:
Thoracoabdominal aneurysm (TAAA) repair is a major elective vascular operation associated with a large blood loss and potentially life-threatening clotting abnormalities. Theses clotting abnormalities are principally treated using fresh frozen plasma (FFP) (derived from human blood donations), the administration of which carries a number of risks including virus transmission (human immunodeficiency virus (HIV), hepatitis B, hepatitis C) and infection with variant Creutzfeld-Jacob disease (vCJD). FFP is no longer administered to children or high-usage adults in the UK because of the infection risk, and recently it was decided by a UK advisory body that the use of UK-derived FFP should cease.

Fibrinogen concentrate is an alternative treatment option to FFP which is thought have less infection risk (purified, heat treated) and has been in licensed use for many years in other European countries. The investigators have been using fibrinogen concentrate recently in their department as an alternative to FFP with encouraging results.

20 patients undergoing elective TAAA repair at The Royal Infirmary of Edinburgh will be randomly allocated to receive standard treatment (FFP) or fibrinogen concentrate as treatment for clotting abnormalities during their surgery. The investigators will take a number of additional blood samples which will provide valuable information about the pattern of clotting abnormalities during this type of operation. The investigators will also record blood loss and the number of allogeneic (derived from human donors) blood components transfused to the patient (red cells, FFP and platelets). Our primary objective is to assess the pattern of coagulation abnormalities in both groups. We will also examine whether the use of fibrinogen concentrate during TAAA repair avoids the need to administer FFP.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective thoracoabdominal aneurysm repair.
* Over 18 years of age.
* Able to give written informed consent.

Exclusion Criteria:

* Previous aortic surgery (re-do surgery).
* Emergency surgery.
* Pregnancy.
* Females of child-bearing age (less than 45 years) not using medically approved method of contraception.
* Congenital or acquired coagulopathy.
* Known allergy to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pattern of coagulation disturbance in the conventional treatment (FFP) and fibrinogen concentrate groups. | Inra-operatively, and up to 24 hours post-operatively.

SECONDARY OUTCOMES:
Proportion of patients in the fibrinogen group in whom FFP transfusion is required during surgery. | Operative period.
Units of FFP transfused - during surgery and up to 24 hours after surgery. | Peri-operative period.
Units of platelets and allogeneic red cells transfused - during surgery and up to 24 hours after surgery. | Peri-operative period.
Blood loss. | Operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Nimmo, MBChB, Principal Investigator — NHS Lothian
Locations (1):
- The Royal Infirmary of Edinburgh, Edinburgh, United Kingdom